CLINICAL TRIAL: NCT05855005
Title: Investigation of Direct-to-consumer Hearing Aids on Conversation Efficiency and Listening Effort
Brief Title: Direct-to-Consumer Hearing Aids and Listening Effort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Pamela Souza, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00217791
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Bilateral
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Bilateral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- DTC Hearing Aid (Experimental)
  Interventions: Device: DTC Hearing Aids

INTERVENTIONS:
Device: DTC Hearing Aids — DTC hearing aid programmed to the individual participant.

SUMMARY:
The aim of this proposed project is to understand whether direct to consumer (DTC) hearing aids programmed to individual hearing losses, can reduce listening effort for effective communication. If DTC aids can provide benefits beyond amplification, then they could be an affordable option to reduce barriers to care and improve hearing aid uptake in adults with hearing loss.

DETAILED DESCRIPTION:
Hearing loss is the third most common chronic health condition in the United States, affecting individuals of any age. According to the National Institute on Deafness and Other Communication Disorders approximately 15% of all adults over age 18 in the United States have reported some trouble with their hearing, and one in eight people in the United States (about 30 million) aged 12 and older have hearing loss in both ears. However, about 28.8 million US adults who could benefit from hearing aids do not wear them. The current model of dispensing hearing aids could be a barrier to adoption by those who could benefit from amplification. Possible barriers from the current model include cost and ability to visit a hearing care professional required to purchase, adjust and repair a hearing aid.

The Food and Drug Administration (FDA) issued a proposal in 2021 to make hearing care more accessible for Americans, known as the Over-the-Counter Hearing Aid Act, part of the FDA Reauthorization Act of 2017. Unlike conventional hearing aids, these devices will not require appointments to an audiologist for adjustments. Due to their affordability and easy access, DTC hearing aids have the potential to reach more individuals with hearing loss. Despite the many potential benefits that DTC hearing aids could offer, there is little research into their use to meet unique patient listening needs and the accuracy of self-guided hearing aid fittings.

The investigators will evaluate the benefit of DTC hearing aids via questionnaires and a conversation task the participant engages in with a familiar speaker.

ELIGIBILITY:
Inclusion Criteria:

1. Speak English as their primary language
2. No vision impairment that would interfere with the ability to complete study tasks (i.e., legally blind, severe cataracts, or macular degeneration)
3. Bilateral mild to moderate sensorineural or mixed hearing loss
4. Pass a cognitive screener
5. Minimum Grade 10 education
6. Ability to attend all study visits
7. Eligible communication partner who can attend first study visit.

Exclusion Criteria:

1. Clinically significant unstable or progressive medical conditions, or conditions which, in the opinion of the investigator(s) places the participant at unacceptable risk if he or she were to participate in the study
2. History of unresolved communication difficulties following another neurological problem (i.e., stroke or brain tumor), neurodevelopmental disorder (i.e., Down's syndrome), or head/neck cancer
3. Diagnosis of dementia or cognitive impairment
4. Positive history of major psychiatric disorder (i.e., schizophrenia, significant untreated depression)
5. Co-enrolled in other intervention studies targeting hearing, language, or communication strategies
6. History or current fluctuating hearing loss
7. Evidence of conductive hearing loss
8. Current active hearing aid wearer (defined as wearing hearing aid(s) at least 4 hours a day for most days within the past year)
9. Current active hearing aid wearer within 30-day trial period of purchased hearing aids from a licensed provider

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Souza, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Chicago, Illinois
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DTC Hearing Aid
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | DTC Hearing Aid
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Diapix Conversation Task: Average Time Per Correctly Identified Difference
Description: Participant and their communication partner discuss pictures with slight differences and attempt to locate all the differences by discussion alone. Primary measurement is average time for each correctly identified difference. A decrease in time indicates improved efficiency in the task.
Time Frame: Task is completed at first study visit (typically 2 hours) after hearing aid fitting, with and without hearing aids.
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | DTC Hearing Aid
Number analyzed (Participants) | 30
Minute
  Unaided | 2.47 (.87)
  Aided | 2.45 (.85)

2. Secondary Outcome: Pupillometry and Recall Repeat Task (RRT)
Description: Participant completes the RRT, a measure of memory and reported listening effort where the listener repeats pre-recorded sentences as they are presented and is then asked to recall them 15 seconds later.
Time Frame: Task will be completed at second study visit (about one hour). second visit usually takes place 1-2 weeks after first visit.
Measure: Mean (Standard Deviation); unit: percentage of words recalled
Arm/Group | DTC Hearing Aid
Number analyzed (Participants) | 30
percentage of words recalled
  Unaided 5 dB SNR Low Context | 23 (12.7)
  Aided (default program per Participant's loss) 5 dB SNR Low Context | 18 (11.12)
  Aided (Noise program) 5 dB SNR Low Context | 21 (12.5)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: This is a non-significant risk study. Participants wore a hearing aid only during their visits to the lab in the presence of the researcher.
Arm/Group | DTC Hearing Aid
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study only used one kind of over the counter hearing aids that only came with a few different levels of amplification. It is possible that a different OTC hearing aid or different patient population would have different outcomes.

The primary outcome measure was also performed in a quiet room with a familiar talker. It is possible that with the same hearing aids but a different task the measured benefit could have been different.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT05855005/Prot_000.pdf